CLINICAL TRIAL: NCT05289011
Title: Spondyloarthritis and Nutrition
Acronym: SANUT
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I17008 (SANUT)
Record Dates: First submitted 2022-03-09; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2020-02

CONDITIONS: Spondyloarthrosis; Nutrition Disorders
Keywords: Spondyloarthrosis; Nutrition Disorders
MeSH Terms: conditions — Spondylarthritis; Nutrition Disorders | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with spondyloarthritis without Inflammatory bowel disease
  Interventions: Other: Interviews and questionnaires

INTERVENTIONS:
Other: Interviews and questionnaires — * Evaluation of inflammatory rheumatism
  * Dietary survey
  * International Physical Activity Questionnaire IPAQ
  * BASDAI self-questionnaire
  * Assessment of quality of life by ASQol questionnaire
  * Assessment of fatigue by FACIT questionnaire
  * Assessment of digestive symptoms
  * Collection of demographic and general data
  * Collection of treatment

SUMMARY:
The food composition and consumption of certain foods could be associated with a higher or lower inflammatory activity of spondyloarthritis and consequently changes in the quality of life of patients. This has been shown in other chronic inflammatory disease.

In order to highlight a profile or nutritional profiles associated with the activity of the disease, we chose to carry out observational pilot study using a qualitative food survey, which will be submitted to all patients with spondyloarthritis. The general demographic data and the data of the disease will be collected by the investigating physician at the same time, as well as possible confounding factors: comorbidities, physical activity, treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who meet the ASAS criteria for axial or peripheral spondyloarthritis
* Patients agreeing to participate and not objecting to the use of their personal data

Exclusion Criteria:

* Presence of Inflammatory bowel disease: Crohn's or RCH diagnosed
* History of bariatric surgery
* Patient subject to a court order, guardianship or trusteeship
* Patient unable to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with axial or peripheral spondyloarthritis
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Nutritional survey | Day 0
  internal questionnaire, correlation between patient's nutrition profile and disease activity
Disease activity | Day 0
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), score ASDAS, correlation between patient's nutrition profile and disease's activity

SECONDARY OUTCOMES:
Physical activity | Day 0
  International Physical Activity Questionnaire (IPAQ)
Assess the quality of life | Day 0
  Ankylosing Spondylitis Quality of Life Questionnaire (ASQol)
Digestive symptoms | Day 0
  Internal questionnaire, correlation between patient's nutrition profile and digestive symptoms The digestive symptom questionnaire had 6 questions, one for each symptom: constipation or hard stools, diarrhoea or frequent stools, stomach pains, gastroesophageal reflux or pyrosis, abdominal pain, and bloating. Each question was scored between 0 to 4: 0 (never occurred), 1 (rarely), 2 (sometimes), 3 (most of the time), and 4 (always). Thus, the cumulative score ranged from 0 to 24
Fatigue | Day 0
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) instrument. The FACIT-F instrument has 13 items with a score ranging from 0 to 52: lower scores indicating more fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No